CLINICAL TRIAL: NCT02113137
Title: Effects of Various Oral Hygiene Procedures on the Reduction of Oral Malodor in Periodontally Healthy Patients
Brief Title: Oral Hygiene Procedures on Reduction of Oral Malodor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ei Ei Aung (Other)
Responsible Party: Sponsor-Investigator, Ei Ei Aung, Graduate student, department of oral health promotion, Tokyo Medical and Dental University
Organization: Tokyo Medical and Dental University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OHP-018-EI
Record Dates: First submitted 2014-04-07; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Halitosis
Keywords: halitosis; chlorine dioxide; tongue cleaning
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1: drug (Experimental): Drug: group 1: drug: chlorine dioxide 12ml chlorine dioxide (ClO2) mouthwash two times per day, for three consecutive weeks
  Interventions: Drug: group 1: drug: chlorine dioxide
- group 2: device: (Experimental): group 2: device: small tooth brush for tongue cleaning small tooth brush for tongue cleaning
  Interventions: Device: group 2: device: small tooth brush for tongue cleaning

INTERVENTIONS:
Drug: group 1: drug: chlorine dioxide — First, each group practiced tooth brushing only for one week. After that each group was requested to do the following procedures.
  group 1 - additional use of 12ml chlorine dioxide (ClO2) mouthwash two times per day, for three consecutive weeks besides tooth brushing.
  At last, each group practiced all three methods of tooth brushing, tongue cleaning, mouth washing.
  Other Names: ClO2Fresh®
  Arms: group 1: drug
Device: group 2: device: small tooth brush for tongue cleaning — First, each group practiced tooth brushing only for one week. After that each group was requested to do the following procedures.
  group 2 - additional practice of tongue cleaning by a small tooth brush two times per day, for three consecutive weeks besides tooth brushing.
  At last, each group practiced all three methods of tooth brushing, tongue cleaning, mouth washing.
  Arms: group 2: device:

SUMMARY:
The purpose of the study is to evaluate the effect of various oral hygiene procedures on reduction of oral malodor.

DETAILED DESCRIPTION:
Thirty volunteers who matched with including criteria were divided randomly into two groups. Both groups were instructed to brush their teeth with a scrubbing method for the first one week. Then, each group received the different additional oral malodor reduction regimen- in addition to tooth brushing tongue cleaning in one group and chlorine dioxide (ClO2) mouthwash in another group for three consecutive weeks. After that, all the participants were instructed to practice all the three oral hygiene procedures (tooth brushing, mouth washing, tongue cleaning) the last one week. Total volatile sulfur compounds (VSCs) measured by breathtron, tongue coating, plaque score and bleeding on probing (BOP) were outcomes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral malodor
* At least 20 functional teeth
* No systemic diseases
* No severe dental diseases

Exclusion Criteria:

* Habit of smoking and betel quid chewing
* Oral malodor by food and other craniofacial abnormalities
* Current use of any kind of mouthwash

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Volatile sulfur compounds (VSCs) | 5 weeks
  Total volatile sulfur compounds was measured by Breathron®

SECONDARY OUTCOMES:
Bleeding on probing | 5 weeks
  gingival bleeding was recorded of bleeding was detected after examination with periodontal probe.
Tongue coating | 5weeks
  tongue coating was evaluated by Winkel tongue coating index.
Debris index | 5 weeks
  debris index was evaluated by oral hygiene index.

CONTACTS AND LOCATIONS:
Overall Officials: EiEi Aung, student, Principal Investigator — Department of oral health promotion
Locations (1):
- Department of oral health promotion, Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Aung EE, Ueno M, Zaitsu T, Furukawa S, Kawaguchi Y. Effectiveness of three oral hygiene regimens on oral malodor reduction: a randomized clinical trial. Trials. 2015 Jan 27;16:31. doi: 10.1186/s13063-015-0549-9. PMID 25622725